CLINICAL TRIAL: NCT06171217
Title: Realizing Effectiveness Across Continents With Hydroxyurea: A Phase I/II Prospective Trial of Hydroxyurea for Children With Sickle Cell Anemia
Brief Title: Realizing Effectiveness Across Continents With Hydroxyurea
Acronym: REACH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-4221b; U01HL133883 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-12-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease; Children
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: The original cohort will continue treatment per planned protocol schedule of evaluations, and a new cohort will join with consent, a 3-month screening period, and treatment per planned protocol schedule of evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Original Cohort (Experimental): The original REACH cohort continuing study treatment per the protocol schedule of evaluations.
  Interventions: Drug: Hydroxyurea
- New Cohort (Experimental): Newly enrolled REACH participants consent, 3 months screening, and treatment per the protocol schedule of evaluations
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea, approximately 20-30 mg/kg/day, with modifications for toxicity or for mild marrow suppression
  Arms: Original Cohort
Drug: Hydroxyurea — Hydroxyurea 15-35 mg/kg/day based on PK-guided dosing, with modifications for toxicity for mild marrow suppression
  Arms: New Cohort

SUMMARY:
REACH is a prospective, phase I/II open-label dose escalation trial of hydroxyurea for children with confirmed SCA between 3 and 10 years of age. The short-term goal is to obtain critical pilot data regarding the feasibility, safety, and benefit of hydroxyurea for children with SCA in multiple distinct research settings in Africa. Based on that information, the longer-term goal is to make hydroxyurea more widely available for children with SCA in Africa, particularly those identified with SCA through expanded newborn screening programs.

DETAILED DESCRIPTION:
REACH is a prospective, phase I/II open-label dose escalation trial of hydroxyurea for children with confirmed SCA between 3 and 10 years of age. The short-term goal is to obtain critical pilot data regarding the feasibility, safety, and benefit of hydroxyurea for children with SCA in multiple distinct research settings in Africa. Based on that information, the longer-term goal is to make hydroxyurea more widely available for children with SCA in Africa, particularly those identified with SCA through expanded newborn screening programs. In the REACH prospective trial, the Original Cohort will receive long-term treatment while for the New Cohort, treatment will continue at least 4 years using PK-guided dosing after an initial 3-month screening period.

ELIGIBILITY:
Inclusion Criteria

1. Pediatric patients with documented sickle cell anemia (typically HbSS supported by hemoglobin electrophoresis, complete blood count, and peripheral blood smear)
2. In the Original Cohort, age range of 1.00-9.99 years, inclusive, at the time of enrollment (now age 5.5 - 17.5 years); age range 3.0-10.0 years for the New Cohort
3. Weight at least 10.0 kg at the time of enrollment
4. Parent or guardian willing and able to provide written informed consent, with child's verbal assent as per local IRB/Ethics Board requirements
5. Willingness to comply with all study-related treatments, evaluations, and follow-up

Exclusion Criteria

1. Known medical condition making participation ill-advised (e.g., acute or chronic infectious disease, HIV, or malignancy)
2. Acute or chronic severe malnutrition determined by impaired growth parameters as defined by WHO (weight for length/height or height for age >3 z-scores below the median WHO growth standards.
3. Pre-existing severe hematological toxicity (temporary exclusions)

   1. Anemia: Hb <4.0 g/dL
   2. Anemia: Hb <6.0 g/dL with ARC <100 x 109/L
   3. Reticulocytopenia: ARC <80 x 109/L with Hb <7.0 g/dL
   4. Thrombocytopenia: Platelets <80 x 109/L
   5. Neutropenia: ANC <1.0 x 109/L
4. Blood transfusion within 60 days before enrollment (temporary exclusion)
5. In the Original Cohort, hydroxyurea use within 6 months before enrollment (temporary exclusion). In the New Cohort, the children should be hydroxyurea naïve, without any prior treatment exposure.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 810 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2027-10-04 (Estimated); Study Completion 2033-10-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of long-term Hydroxyurea treatment at MTD | Assessed every 6 ± 1 months up to 204 months
  The efficacy of hydroxyurea will be primarily assessed through fetal hemoglobin (HbF), comparing treatment with baseline values.

SECONDARY OUTCOMES:
Reduction of malaria incidents while on hydroxyurea at MTD. | Assessed every 4 ± 1 weeks, then every 3 ± 1months up to 204 months
  Clinical malaria infections to identify associations of risk or protection comparing treated and untreated incidents.
Success of PK-guided dosing of hydroxyurea | Assessed every 6 ± 1 months up to 204 months
  Fetal Hemoglobin changes from hydroxyurea at MTD

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- Hospital Pediátrico David Bernardino, Luanda, Angola
- Centre Hospitalier Monkole, Kinshasa, Democratic Republic of the Congo
- KEMRI/Wellcome Trust Research, Kilifi, Kenya
- Mbale Regional Hospital, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Investigators whose proposed use of the data has been approved by a review committee identified for this purpose, will be provided individual participant data that underlie the results reported from this study, after de-identification and publication. The data can be obtained via email to Dr. Ware as the corresponding author.
Supporting Information: Study Protocol
Time Frame: Nine months following publication ending 36 months following publication.
Access Criteria: For individual participant data meta-analysis after approval of a proposal and with a signed data access agreement.